CLINICAL TRIAL: NCT00296374
Title: Randomised, Double-blind, 52-wk, Parallel-grp, Multicentre, PIIb Study to Evaluate Effects of Rosuvastatin 10mg, Rosuvastatin 40mg and Atorvastatin 80mg on Urinary Protein Excretion in Hypercholesterolaemic Diabetic Patients With Moderate Proteinuria
Brief Title: Prospective Evaluation of Proteinuria and Renal Function in Diabetic Patients With Progressive Renal Disease
Acronym: PLANET 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3569C00007; PLANET 1
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus
Keywords: Hyperlipidemia; Proteinuria; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Proteinuria | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Rosuvastatin 10 mg
  Interventions: Drug: Rosuvastatin
- 2 (Experimental): Rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin
- 3 (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg oral dose administered once daily for 52 weeks
  Other Names: Crestor
  Arms: 1
Drug: Rosuvastatin — 20 mg oral dose administered once daily for 4 weeks followed by 40 mg oral dose administered once daily for 48 weeks
  Other Names: Crestor
  Arms: 2
Drug: Atorvastatin — 40 mg oral dose administered once daily for 4 weeks followed by 80 mg oral dose administered once daily for 48 weeks
  Other Names: Lipitor
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effects of Crestor (rosuvastatin) and (Lipitor) atorvastatin on urinary protein excretion over 1 year in patients with Type 1 or 2 diabetes with moderate proteinuria and hypercholesterolaemia.

ELIGIBILITY:
Inclusion Criteria:

* hyperlipidemia
* urinary protein
* diabetes

Exclusion Criteria:

* previous rosuvastatin treatment < 6 months prior to Visit 1
* statin intolerance
* severe hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Science Director, MD, Study Director — AstraZeneca
Locations (116):
- United States (29):
  - Research Site, Avondale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Pasadena, California
  - Research Site, Riverside, California
  - Research Site, Santa Ana, California
  - Research Site, West Hills, California
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Topeka, Kansas
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Orchard Park, New York
  - Research Site, Stony Brook, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
  - Research Site, Milwaukee, Wisconsin
- Argentina (4):
  - Research Site, Buenos Aires
  - Reasearch Site, La Plata
  - Research Site, Morón
  - Research Site, Quilmes
- Brazil (5):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Recife
  - Research Site, São Paulo
- Bulgaria (7):
  - Research Site, Burgas
  - Research Site, Gabrovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Courtice, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Blegdamsvej 9
  - Research Site, Farsø
  - Research Site, Gentofte Municipality
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, Køge
- France (13):
  - Research Site, Annonay
  - Research Site, Besançon
  - Research Site, Bondy
  - Research Site, Colmar
  - Research Site, Corbeil-Essonnes
  - Research Site, Corsept
  - Research Site, Creil
  - Research Site, Grenoble
  - Research Site, La Chapelle-sur-Erdre
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Quimper
- Hungary (16):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research site, Gyula
  - Research Site, Hodmeztvasarhely
  - Research Site, Kecskemét
  - Research Site, Keszthely
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Tatabánya
  - Research Site, Zalaegerszeg
- Italy (10):
  - Research Site, Acireale, CT
  - Research Site, Florence, FI
  - Research Site, Roma, RM
  - Research Site, Sottomarnia Di Chioggia, VE
  - Research Site, Bergamo
  - Research Site, Cagliari
  - Research Site, Milan
  - Research Site, San Giovanni Rotondo
  - Research Site, Sassari
  - Research Site, Treviglio
- Mexico (8):
  - Research Site, Aguascalientes
  - Research Site, Cauntla
  - Research Site, Distrito Federal
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Saltillo
  - Research Site, San Luis Potosí City
  - Research Site, Zapopan
- Romania (7):
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Lasi
  - Research Site, Târgu Mureş
  - Research Site, Timișoara

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] de Zeeuw D, Anzalone DA, Cain VA, Cressman MD, Heerspink HJ, Molitoris BA, Monyak JT, Parving HH, Remuzzi G, Sowers JR, Vidt DG. Renal effects of atorvastatin and rosuvastatin in patients with diabetes who have progressive renal disease (PLANET I): a randomised clinical trial. Lancet Diabetes Endocrinol. 2015 Mar;3(3):181-90. doi: 10.1016/S2213-8587(14)70246-3. Epub 2015 Feb 4. PMID 25660356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 353 patients entered the study with Type 1 or 2 diabetes and were receiving current treatment with angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blockers (ARBs). The study was conducted at 147 centers in 11 countries.
Pre-assignment Details: Patients requiring an adjustment of the ACE inhibitor and/or ARBs after Visit 1 were excluded. All 353 patients were randomized and 276 patients completed the study.
Period: Overall Study
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Started | 118 | 124 | 111
Completed | 93 | 101 | 82
Not Completed | 25 | 23 | 29
Not completed — Adverse Event | 14 | 10 | 7
Not completed — Withdrawal by Subject | 3 | 5 | 11
Not completed — Incorrect enrollment | 3 | 3 | 4
Not completed — Protocol Violation | 1 | 2 | 3
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Relocated to another state | 1 | 0 | 0
Not completed — Stopped drug before end of study visit | 0 | 1 | 0
Not completed — Nephrologist introduced ACE | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg | Total
Number analyzed (Participants) | 118 | 124 | 111 | 353
Age, Customized [Number; unit: Participants]
  18-49 years | 22 | 33 | 25 | 80
  50-64 years | 59 | 59 | 57 | 175
  >=65 years | 37 | 32 | 29 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 32 | 33 | 108
  Male | 75 | 92 | 78 | 245
Estimated glomerular filtration rate [eGFR] [Mean (Standard Deviation); unit: mL/min] | 68.759 (24.1080) | 72.644 (25.8018) | 72.149 (24.8721) | 71.210 (24.9455)
Urine albumin/creatinine ratio [Mean (Standard Deviation); unit: mg/g] | 1036.478 (730.6185) | 1079.802 (725.7039) | 1143.198 (779.5282) | 1085.435 (743.5360)
Urine protein/creatinine ratio [Mean (Standard Deviation); unit: mg/g] | 1392.26 (888.3215) | 1493.574 (996.0972) | 1517.858 (969.7020) | 1467.843 (952.0380)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Protein/Creatinine Ratio in Patients With Type 1 or 2 Diabetes.
Description: Urinary protein/creatinine ratio (mg/g) =urine protein concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 52 [LOCF] urine protein/creatinine ratio over baseline urine protein/creatinine ratio.
Time Frame: Assessed at Week 52, Last observation carried forward (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Number analyzed (Participants) | 107 | 116 | 102
mg/g | 1.016 [0.858 to 1.209] | 0.955 [0.869 to 1.185] | 0.874 [0.733 to 0.975]

2. Secondary Outcome: Urinary Protein/Creatinine Ratio at Week 26.
Description: Urinary protein/creatinine ratio (mg/g) =urine protein concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 26 urine protein/creatinine ratio over baseline urine protein/creatinine ratio.
Time Frame: Assessed at Week 26
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Number analyzed (Participants) | 98 | 108 | 92
mg/g | 1.007 [0.895 to 1.133] | 0.994 [0.881 to 1.121] | 0.876 [0.784 to 0.979]

3. Secondary Outcome: Urinary Albumin/Creatinine Ratio at Week 26
Description: Urinary albumin/creatinine ratio (mg/g) =urine albumin concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 26 urine albumin/creatinine ratio over baseline urine albumin/creatinine ratio.
Time Frame: Assessed at Week 26
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Number analyzed (Participants) | 98 | 109 | 92
mg/g | 0.927 [0.792 to 1.085] | 0.913 [0.788 to 1.058] | 0.831 [0.726 to 0.951]

4. Secondary Outcome: Urinary Albumin/Creatinine Ratio at Week 52 [LOCF]
Description: Urinary albumin/creatinine ratio (mg/g) =urine albumin concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 52 [LOCF] urine albumin/creatinine ratio over baseline urine albumin/creatinine ratio.
Time Frame: Assessed at Week 52 LOCF
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Number analyzed (Participants) | 107 | 116 | 102
mg/g | 1.016 [0.856 to 1.206] | 0.836 [0.704 to 0.993] | 0.823 [0.709 to 0.954]

5. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 26
Time Frame: Assessed at Baseline and Week 26
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Number analyzed (Participants) | 100 | 111 | 92
mL/min | -2.73 (12.644) | -5.46 (14.079) | -1.78 (10.997)

6. Secondary Outcome: Change From Baseline in eGFR at Week 52 [LOCF]
Time Frame: Assessed at Baseline and Week 52 [LOCF]
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 107 | 115 | 101
mL/min | -3.70 (14.551) | -7.29 (20.040) | -1.61 (12.769)

7. Secondary Outcome: Correlation Coefficient Urinary Protein/Creatinine Ratio and Total Cholesterol [TC] Indicating the Relationship Between Renal Effects and Lipid Changes
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 52 (LOCF).
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Groups:
- Rosuvastatin: Rosuvastatin Treatments pooled
- Atorvastatin: Atorvastatin Treatment
- All Treatment: All Treatments pooled
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 205 | 91 | 296
Correlation coefficient | -0.03507 | 0.14258 | 0.01600

8. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio TC
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 52
Time Frame: Assessed at 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 79 | 269
Correlation coefficient | 0.07019 | 0.26855 | 0.12013

9. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and Low Density Lipoprotein Cholesterol [LDL-C]
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 26.
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | -0.08588 | 0.18570 | -0.02491

10. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and LDL-C
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | 0.04510 | 0.16280 | 0.06739

11. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and High Density Lipoprotein Cholesterol [HDL-C]
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | 0.15614 | 0.06987 | 0.14226

12. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and HDL-C
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | 0.16111 | 0.26194 | 0.18918

13. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and Non-high Density Lipoprotein Cholesterol [nonHDL-C]
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | -0.12068 | 0.15929 | -0.05186

14. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and nonHDL-C
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | 0.02594 | 0.24018 | 0.07381

15. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and Triglyceride [TG]
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 205 | 91 | 296
Correlation coefficient | -0.14569 | 0.04948 | -0.08471

16. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and TG
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 269
Correlation coefficient | -0.05251 | 0.11755 | 0.01345

17. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and TC/HDL-C Ratio
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | -0.13572 | 0.07339 | -0.08855

18. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and TC/HDL-C Ratio
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | -0.05945 | 0.12132 | -0.02666

19. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and LDL-C/HDL-C Ratio
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | -0.13689 | 0.12931 | -0.08108

20. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and LDL-C/HDL-C Ratio
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | -0.02775 | 0.06535 | -0.01569

21. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and nonHDL-C/HDL-C Ratio
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 203 | 90 | 293
Correlation coefficient | -0.16755 | 0.08891 | -0.11221

22. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and nonHDL-C/HDL-C Ratio
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 190 | 78 | 268
Correlation coefficient | -0.06085 | 0.12507 | -0.02841

23. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and Apolipoprotein A-1 [ApoA-1]
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 87 | 278
Correlation coefficient | 0.15859 | 0.13133 | 0.15516

24. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and ApoA-1
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 183 | 78 | 261
Correlation coefficient | 0.16587 | 0.18469 | 0.18832

25. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and Apolipoprotein B [ApoB]
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 87 | 278
Correlation coefficient | -0.02276 | 0.21405 | 0.04578

26. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and ApoB
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 183 | 78 | 261
Correlation coefficient | 0.05397 | 0.29486 | 0.11079

27. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and ApoB/ApoA-1 Ratio
Description: as for outcome 9
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 87 | 278
Correlation coefficient | -0.07846 | 0.13910 | -0.02825

28. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Protein/Creatinine Ratio and ApoB/ApoA-1 Ratio
Description: as for outcome 8
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 183 | 78 | 261
Correlation coefficient | 0.00600 | 0.22710 | 0.03684

29. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TC
Description: Correlation of changes from baseline in urinary albumin/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 26.
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 206 | 91 | 297
Correlation coefficient | 0.00642 | 0.14331 | 0.04311

30. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TC
Description: Correlation of changes from baseline in urinary albumin/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 52
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 79 | 270
Correlation coefficient | 0.13220 | 0.35715 | 0.18971

31. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and LDL-C
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | -0.05514 | 0.19842 | 0.00038

32. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and LDL-C
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.10037 | 0.21205 | 0.12270

33. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and HDL-C
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | 0.08593 | 0.00032 | 0.06930

34. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and HDL-C
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.14758 | 0.26805 | 0.17550

35. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and nonHDL-C
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | -0.06694 | 0.17296 | -0.01144

36. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and nonHDL-C
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.09189 | 0.33769 | 0.14988

37. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TG
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 206 | 91 | 297
Correlation coefficient | -0.07271 | 0.08654 | -0.02876

38. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TG
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 79 | 270
Correlation coefficient | -0.02947 | 0.27198 | 0.08787

39. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TC/HDL-C Ratio
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | -0.04785 | 0.11256 | -0.01362

40. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and TC/HDL-C Ratio
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.01798 | 0.20127 | 0.05369

41. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and LDL-C/HDL-C Ratio
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | -0.08211 | 0.16654 | -0.03001

42. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and LDL-C/HDL-C Ratio
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.03476 | 0.10902 | 0.04508

43. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and nonHDL-C/HDL-C Ratio
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 204 | 90 | 294
Correlation coefficient | -0.08468 | 0.12805 | -0.04102

44. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and nonHDL-C/HDL-C Ratio
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 191 | 78 | 269
Correlation coefficient | 0.01528 | 0.21198 | 0.05251

45. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoA-1
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 192 | 87 | 279
Correlation coefficient | 0.14207 | 0.11171 | 0.13429

46. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoA-1
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 184 | 78 | 262
Correlation coefficient | 0.16085 | 0.15933 | 0.17306

47. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoB
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 192 | 87 | 279
Correlation coefficient | -0.00569 | 0.20008 | 0.04833

48. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoB
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 184 | 78 | 262
Correlation coefficient | 0.10997 | 0.30537 | 0.15652

49. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoB/ApoA-1 Ratio
Description: as for outcome 29
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 192 | 87 | 279
Correlation coefficient | -0.05906 | 0.13706 | -0.01775

50. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: Urinary Albumin/Creatinine Ratio and ApoB/ApoA-1 Ratio
Description: as for outcome 30
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 184 | 78 | 262
Correlation coefficient | 0.04760 | 0.25636 | 0.07766

51. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TC
Description: Correlation of changes from baseline in eGFR with percent change from baseline in lipids and lipoprotein concentrations at Week 26.
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 211 | 91 | 302
Correlation coefficient | 0.01586 | -0.03124 | 0.00101

52. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TC
Description: Correlation of changes from baseline in eGFR with percent change from baseline in lipids and lipoprotein concentrations at Week 52
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 82 | 277
Correlation coefficient | -0.13489 | -0.18105 | -0.14690

53. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and LDL-C
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | 0.03010 | -0.00944 | 0.02609

54. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and LDL-C
Description: as for outcome 52
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | -0.11072 | -0.12835 | -0.11378

55. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and HDL-C
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | 0.11373 | 0.01123 | 0.07576

56. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and HDL-C
Description: as for outcome 52
Time Frame: 52 Weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | 0.14457 | -0.15546 | 0.08841

57. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and nonHDL-C
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | -0.01709 | -0.05610 | -0.02569

58. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and nonHDL-C
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | -0.17729 | -0.19501 | -0.17911

59. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TG
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 211 | 91 | 302
Correlation coefficient | -0.10533 | -0.00604 | -0.09437

60. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TG
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 82 | 277
Correlation coefficient | -0.24494 | -0.07059 | -0.15586

61. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TC/HDL-C Ratio
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | -0.05426 | -0.01643 | -0.04256

62. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and TC/HDL-C Ratio
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | -0.26268 | -0.08593 | -0.23226

63. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and LDL-C/HDL-C Ratio
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | -0.01040 | 0.00241 | 0.00189

64. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and LDL-C/HDL-C Ratio
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | -0.19850 | -0.06481 | -0.17579

65. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and nonHDL-C/HDL-C Ratio
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 209 | 90 | 299
Correlation coefficient | -0.06356 | -0.04402 | -0.05499

66. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and nonHDL-C/HDL-C Ratio
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 195 | 81 | 276
Correlation coefficient | -0.26802 | -0.11804 | -0.24204

67. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoA1
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 197 | 87 | 284
Correlation coefficient | 0.08146 | 0.05333 | 0.05845

68. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoA1
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 187 | 81 | 268
Correlation coefficient | 0.17909 | 0.08090 | 0.12787

69. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoB
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 197 | 87 | 284
Correlation coefficient | -0.01427 | 0.08821 | 0.00737

70. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoB
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 187 | 81 | 268
Correlation coefficient | -0.15146 | 0.04886 | -0.12168

71. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoB/ApoA-1 Ratio
Description: as for outcome 51
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 197 | 87 | 284
Correlation coefficient | -0.04088 | 0.06598 | -0.01652

72. Secondary Outcome: Relationship Between Renal Effects and Lipid Changes: eGFR and ApoB/ApoA-1 Ratio
Description: as for outcome 52
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatment
Number analyzed (Participants) | 187 | 81 | 268
Correlation coefficient | -0.26146 | 0.05248 | -0.22109

ADVERSE EVENTS:
Arm/Group | Rosuvastatin 10mg | Rosuvastatin 40mg | Atorvastatin 80mg
Serious Adverse Events (participants affected / at risk) | 18/116 | 20/123 | 21/110
Other Adverse Events (participants affected / at risk) | 15/116 | 25/123 | 12/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10mg (N=116) | Rosuvastatin 40mg (N=123) | Atorvastatin 80mg (N=110)
Cardiac Failure (Cardiac disorders) | 3 | 1 | 1
Angina Pectoris (Cardiac disorders) | 2 | 1 | 2
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Diabetic Eye Disease (Eye disorders) | 1 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0 | 0
Diabetic Retinopathy (Eye disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 2 | 0 | 0
Death (General disorders) | 1 | 1 | 0
Soft Tissue Inflammation (General disorders) | 1 | 0 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 1 | 0 | 0
Abdominal Infection (Infections and infestations) | 0 | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Factitious Disorder (Psychiatric disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 2 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Femoral Arterial Stenosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Poor Peripheral Circulation (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10mg (N=116) | Rosuvastatin 40mg (N=123) | Atorvastatin 80mg (N=110)
Oedema Peripheral (General disorders) | 9 | 5 | 3
Influenza (Infections and infestations) | 3 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 7
Hypertension (Vascular disorders) | 2 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less